CLINICAL TRIAL: NCT02543541
Title: A Pilot Study of Structured Palliative Care for Patients Enrolled on Phase I Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5Y15
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Cancer
Keywords: Palliative Care; Supportive Care; Caregiver; Phase I
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Supportive Care (Active Comparator)
  Interventions: Behavioral: Standard supportive care
- Structured Supportive Care (Experimental)
  Interventions: Behavioral: Structured palliative care

INTERVENTIONS:
Behavioral: Structured palliative care — Supportive care for the patient and caregiver will be provided by the outpatient palliative care team which includes clinicians with specialized palliative care training, social workers, spiritual care specialists and mental health clinical nurse specialist.
  Arms: Structured Supportive Care
Behavioral: Standard supportive care — Supportive care for the patient and caregiver will be provided by the treating oncologist.
  Arms: Standard Supportive Care

SUMMARY:
The goal of this research study is to find out if providing patients who are enrolled in phase 1 clinical trials with structured supportive care will enable them to continue in the Phase 1 trial longer and improve their quality of life by reducing or treating side effects and by providing emotional and social support to the patient and family. The structured supportive or palliative care intervention will be provided by a team of trained specialists which include doctors, nurses, social workers and spiritual care providers. The supportive care team will provide treatment to address symptoms, such as pain or anxiety, caused by the cancer itself or from the treatment. The team can make referrals to other specialists. Such as psychologists or nutritionist, if needed, and can help arrange for services to address home care needs.

DETAILED DESCRIPTION:
Primary Objective(s): To assess symptoms, adverse events, duration on study, reason for study discontinuation, and quality of life among patients participating in phase I clinical trials who receive structured palliative care, and those who receive standard supportive care. Duration on study will serve as the primary objective for sample size determination.

Secondary Objective(s):

1. To describe the quantity (e.g. hours), type, and cost of palliative care personnel services used by patients and caregivers receiving structured palliative care.

Exploratory:

1. To compare adverse event profiles, duration on study, and quality of life between patients who receive structured palliative care and those receiving standard supportive care.
2. To compare caregiver burden and quality of life between the study arms.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patients must be enrolled in a Phase 1 clinical trial and be within 2 weeks of starting the experimental therapy or intervention.
* Patients are eligible to enroll on this study with or without the enrollment of their caregiver.

Patient Exclusion Criteria:

* Patients diagnosed with a hematologic malignancy.

Caregiver Inclusion Criteria:

* Any caregiver is considered eligible for this study; The caregiver is the person identified by the patient as the one who provides the most regular physical and/or emotional support.
* Caregivers must be willing to complete surveys at baseline and on monthly basis.

Caregiver Exclusion Criteria:

* Caregivers who are solely professional, paid caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-10-25; Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Average total MSAS score | Up to 6 months
  Assessment of patient burden
Average total FACT-G score | Up to 6 months
  Measure patient quality of life
Reason for study discontinuation (Patient reported outcome) | Up to 6 months
  Measure of central tendency for why patients discontinued the phase I study. Patient reported outcomes for reason for study discontinuation will be qualitatively assessed
Duration on Study | Up to 6 months
  Measure of central tendency of the duration patients were on the phase I study. Duration on study will serve as the primary objective for sample size determination
Adverse events | Up to 6 months
  Measure of central tendency of adverse events. AE will be described and further categorized as modifiable (primary symptom experience) and non-modifiable (laboratory abnormalities). The influence of adverse events on study outcomes particularly duration on study and reason for study discontinuation will be assessed. An exploratory weighted adverse event score will be calculated using the equation: adverse event score = ∑ (NAE * GAE) where N denotes the adverse event number, G denotes grade, AE denotes adverse event. These scores will be compared between study arms

SECONDARY OUTCOMES:
Mean number of hours of palliative care services | Up to 6 months
  Mean number of hours utilized by patients and caregivers who received structured palliative care. This analysis will be descriptive, reporting measures of central tendency
Type of palliative care services | Up to 6 months
  Measure of central tendency for the type of palliative care services utilized by patients and caregivers who received structured palliative care. This analysis will be descriptive, reporting measures of central tendency

OTHER OUTCOMES:
Frequency of adverse events of patients receiving structured and usual supportive care | Up to 6 months
Average days on study | Up to 6 months
Change in FACT-G score | From baseline to last contact, up to 6 months
  Change in patient symptom burden when compared to baseline between patients who received structured palliative care and those who received standard supportive care
Change in MSAS score | From baseline to last contact, up to 6 months
  Change in quality of life when compared to baseline between patients who received structured palliative care and those who received standard supportive care
Change in CRA score | From baseline to last contact, up to 6 months
  Change in caregiver burden when compared to baseline between those who received structured palliative care and those who received standard supportive care
Change in QOLLTI-F score | From baseline to last contact, up to 6 months
  Change in caregiver quality of life as assessed through change in QOLLTI-F score when compared to baseline between those who received structured palliative care and those who received standard supportive care

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Treasure, MD, Principal Investigator — Metrohealth Medical Center and Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Treasure M, Daly B, Cao S, Fu P, Hong A, Weinstein E, Surdam J, Meropol NJ, Dowlati A. A randomized controlled trial of structured palliative care versus standard supportive care for patients enrolled in phase 1 clinical trials. Cancer Med. 2021 Jul;10(13):4312-4321. doi: 10.1002/cam4.3971. Epub 2021 May 25. PMID 34033228